CLINICAL TRIAL: NCT03015883
Title: A Safety and Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters on Squamous Cell Carcinoma (First in Man)
Brief Title: Alpha Radiation Emitters Device for the Treatment of Squamous Cell Carcinoma
Acronym: DaRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-SCC-00
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma; Alpha emitting radiation; Skin Cancer; Carcinoma, Squamous; HNSCC
MeSH Terms: conditions — Carcinoma, Squamous Cell; Skin Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diffusing Alpha Radiation Emitters Therapy (DaRT) (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seed Devices
  Interventions: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.
  Other Names: DaRT

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device.

DETAILED DESCRIPTION:
This will be a prospective, first in man, controlled study, assessing the safety and efficacy of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Lesions with histopathological diagnosis of squamous cell carcinoma will be studied.

Reduction in tumor size 30 days after DaRT insertion will be assessed.

Safety will be assessed by the incidence, severity and frequency of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological confirmation of squamous cell carcinoma.
2. Tumor size ≤ 5 centimeters in the longest diameter.
3. Age over 18.
4. Women of childbearing potential will have evidence of negative pregnancy test.
5. Life expectancy of more than 6 months.
6. Performance status 2 (ECOG scale) or less.
7. Signed informed consent form.

Exclusion Criteria:

1. Tumor maximal diameter > 5 centimeters.
2. Tumor of Keratoacanthoma histology.
3. Performance status ≥ 3 (ECOG scale).
4. Patients with moribund diseases, autoimmune diseases or vasculitis.
5. Patients under immunosuppressive and/or corticosteroid treatment.
6. Volunteers that participated in other studies in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30-45 days post seed insertion
  The incidence, severity and frequency of all Adverse Events
Reduction in Tumor size | 30-45 days post seed insertion
  The reduction in tumor size 30-45 days after DaRT insertion

SECONDARY OUTCOMES:
Percent of NecroticTissue | 30-45 days post seed insertion
  Percent of necrotic tissue in the tumor 30 days after DaRT insertion

CONTACTS AND LOCATIONS:
Overall Officials: Noga Kurman, MD, Principal Investigator — Davidof Cancer Institution at the Rabin Medical Center Israel
Locations (1):
- Davidof Cancer Institution at the Rabin Medical Center Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No